CLINICAL TRIAL: NCT05138549
Title: Effect of Astaxanthin for Pain, Function, and Inflammation in Patients With Advanced Osteoarthritis Awaiting Total Knee Replacement Surgery
Brief Title: Astaxanthin for Management of Inflammation in Knee Osteoarthritis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: There are not enough eligible patients at our institution to complete this study.
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00113612
Record Dates: First submitted 2021-10-28; First posted 2021-12-01 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis Knees Both; Joint Inflammation
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive 6 weeks of oral supplementation of either placebo or 12 mg astaxanthin prior to total knee replacement surgery.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers, and investigators will not know which arm patients have been assigned to or if they receive placebo or astaxanthin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control: Placebo Group (Placebo Comparator): Patients will receive a 6 week daily oral supply of placebo, identical in appearance to the astaxanthin supplement.
  Interventions: Other: Placebo
- Experimental: Astaxanthin Supplementation Group (Active Comparator): Patients will receive a 6 week daily oral supply of 12 mg astaxanthin supplement.
  Interventions: Drug: Astaxanthin

INTERVENTIONS:
Drug: Astaxanthin — 12 mg oral astaxanthin supplement
  Other Names: Astaxanthine; Astaxantina; Dihydroxy-3,3' dioxo-4,4' bêta-carotène
  Arms: Experimental: Astaxanthin Supplementation Group
Other: Placebo — Oral placebo identical to astaxanthin supplement
  Arms: Control: Placebo Group

SUMMARY:
Over 30 million Americans are currently affected by osteoarthritis (OA), with prevalence expected to increase 40% by 2025 as a result of the aging population and obesity epidemic. Specifically, symptomatic knee OA is a leading cause of disability. Although originally classified as non-inflammatory arthritis, recent studies suggest that a relationship exists between joint inflammation and OA. Specifically, the complex interaction between sites of local tissue damage and immune cells leads to a state of chronic joint inflammation which may play a key role in disease pathogenesis. The evidence suggesting a role of inflammation in disease progression makes anti-inflammatory agents ideal candidates for symptom management. Astaxanthin, a keto-carotenoid present in many aquatic animals, including salmon, shrimp, and lobster, is an FDA-approved nutraceutical that has powerful antioxidant and anti-inflammatory properties coupled with remarkable safety and tolerability. This prospective, blinded, randomized, placebo-controlled pilot study will evaluate the effect of astaxanthin in reducing inflammation, controlling pain, and improving physical function in patients with advanced knee osteoarthritis awaiting total joint replacement surgery. Levels of pro- and anti-inflammatory cytokines and chemokines will be measured following the completion of a daily oral regimen of astaxanthin vs. placebo. Additionally, patient-reported outcome measurements assessing physical function and pain interference will be obtained prior to and following completion of treatment allowing for a comparison between treatment groups. Study outcomes will provide evidence to support astaxanthin supplementation as a cost-effective, added strategy for symptom management in patients with advanced osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common degenerative joint disorder that affects a significant portion of the population. Over 30 million Americans are currently affected by the disease, with prevalence expected to increase 40% by 2025 as a result of the aging population and obesity epidemic. Specifically, symptomatic knee OA is a leading cause of disability, occurring in 10% of men and 13% of women over the age of 60. Patients with symptomatic OA often experience pain, swelling, and stiffness of the knee resulting in a decrease in physical mobility which can have a drastic impact on quality of life. In addition to the significant impact on affected individuals, OA is associated with an enormous economic burden estimated at $136.8 billion annually in the US, surpassing costs of tobacco-related health effects, diabetes, and cancer.

Although originally classified as non-inflammatory arthritis, recent studies suggest that a relationship exists between joint inflammation and OA. Specifically, the complex interaction between sites of local tissue damage and immune cells leads to a state of chronic joint inflammation which may play a key role in disease pathogenesis. The evidence suggesting a role of inflammation in disease progression makes anti-inflammatory agents ideal candidates for symptom management. Astaxanthin is a keto-carotenoid present in many aquatic animals, including salmon, shrimp, and lobster, that has demonstrated heightened antioxidant activity and the ability to suppress inflammation. Early evidence suggests that astaxanthin may protect against osteoarthritis in vivo, illustrating its potential as a therapeutic supplement for patients with OA. However, studies illustrating these effects in humans have yet to be conducted.

This prospective, blinded, randomized, placebo-controlled pilot study will evaluate the effect of astaxanthin in reducing inflammation, controlling pain, and improving physical function in patients with advanced knee osteoarthritis awaiting total joint replacement surgery. Levels of pro- and anti-inflammatory cytokines and chemokines will be measured following the completion of a daily oral regimen of astaxanthin vs. placebo. Additionally, patient-reported outcome measurements assessing physical function and pain interference will be obtained prior to and following completion of treatment allowing for a comparison between treatment groups. Study outcomes will provide evidence to support astaxanthin supplementation as a cost-effective, added strategy for symptom management in patients with advanced osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Radiographic evidence of advanced knee osteoarthritis
* Knee pain
* Scheduled to undergo a total knee replacement

Exclusion Criteria:

* < 18 years of age
* Unable to provide written consent
* Known allergy to fish or astaxanthin
* Pregnant and/or breastfeeding
* Received a corticosteroid injection within 3 months of initiating treatment with astaxanthin or placebo
* Currently taking immunosuppressants
* Patients with known autoimmune etiology for arthritis (e.g. Rheumatoid or Psoriatic arthritis)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Del Gaizo, MD, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Prisma Health, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Sun K, Luo J, Jing X, Guo J, Yao X, Hao X, Ye Y, Liang S, Lin J, Wang G, Guo F. Astaxanthin protects against osteoarthritis via Nrf2: a guardian of cartilage homeostasis. Aging (Albany NY). 2019 Nov 26;11(22):10513-10531. doi: 10.18632/aging.102474. Epub 2019 Nov 26. PMID 31772142
- [Background] Farr Ii J, Miller LE, Block JE. Quality of life in patients with knee osteoarthritis: a commentary on nonsurgical and surgical treatments. Open Orthop J. 2013 Nov 13;7:619-23. doi: 10.2174/1874325001307010619. eCollection 2013. PMID 24285987
- [Background] Vitaloni M, Botto-van Bemden A, Sciortino Contreras RM, Scotton D, Bibas M, Quintero M, Monfort J, Carne X, de Abajo F, Oswald E, Cabot MR, Matucci M, du Souich P, Moller I, Eakin G, Verges J. Global management of patients with knee osteoarthritis begins with quality of life assessment: a systematic review. BMC Musculoskelet Disord. 2019 Oct 27;20(1):493. doi: 10.1186/s12891-019-2895-3. PMID 31656197
- [Background] Sokolove J, Lepus CM. Role of inflammation in the pathogenesis of osteoarthritis: latest findings and interpretations. Ther Adv Musculoskelet Dis. 2013 Apr;5(2):77-94. doi: 10.1177/1759720X12467868. PMID 23641259
- [Background] Scanzello CR, Goldring SR. The role of synovitis in osteoarthritis pathogenesis. Bone. 2012 Aug;51(2):249-57. doi: 10.1016/j.bone.2012.02.012. Epub 2012 Feb 22. PMID 22387238
- [Background] Higuera-Ciapara I, Felix-Valenzuela L, Goycoolea FM. Astaxanthin: a review of its chemistry and applications. Crit Rev Food Sci Nutr. 2006;46(2):185-96. doi: 10.1080/10408690590957188. PMID 16431409
- [Background] Park JS, Chyun JH, Kim YK, Line LL, Chew BP. Astaxanthin decreased oxidative stress and inflammation and enhanced immune response in humans. Nutr Metab (Lond). 2010 Mar 5;7:18. doi: 10.1186/1743-7075-7-18. PMID 20205737

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group
Started | 10 | 6
Completed | 5 | 4
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12.4) | 74 (10.7) | 69 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 5 | 6 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Effect of Astaxanthin on Inflammatory Synovial Markers in Patients With Osteoarthritis Who Are Scheduled to Undergo a Total Knee Replacement Surgery.
Description: We will address this by conducting a prospective, double-blinded, randomized, placebo-controlled trial in which 160 patients who have been diagnosed with advanced osteoarthritis of the knee and are scheduled to undergo a total knee replacement will randomly receive a 6-week oral daily course of either astaxanthin (12 mg) or placebo prior to surgery. Levels of pro- and anti-inflammatory cytokines and chemokines within the intra-articular synovial fluid at the time of surgery will be quantified using a bioplex 23-cytokine and chemokine assay kit in post-treatment synovial fluid samples from patients receiving either astaxanthin or placebo.
Time Frame: 6 Weeks
Population: The synovial fluid samples were being held to be batch processed at the end of the study by an outside scientific laboratory. The study was stopped early and the cytokine and chemokines testing was not done. There are no plans to analyze these samples at present or in the future. Therefore, there are no results to report for this outcome measure which is why participants analyzed for the control and experimental groups are both 0.
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Effect of Astaxanthin on PROMIS Physical Function Scores in Patients With Osteoarthritis Who Are Scheduled to Undergo a Total Knee Replacement Surgery.
Description: Patient reported outcomes will be collected utilizing the Patient Reported Outcome Measurement Information Systems (PROMIS) Physical Function assessment tool. Patients receiving either astaxanthin or placebo will complete PROMIS Physical Function assessment prior to starting the oral treatment regimen and just prior to surgery, following the completion of the oral treatment regimen. As the PROMIS tool has national normative data for age, sex, and condition, collection of patient-reported outcomes in this manner will allow for comparison between patients receiving astaxanthin and patients receiving the placebo as well as the general population. An increased PROMIS Physical Function score indicates an improvement in patient-reported physical function. The scale range is 0 to 100 with a mean of 50 and a standard deviation of 10. Higher values are associated with more or higher function. A score of 60 is one SD better than average. A score of 40 is one SD worse than average.
Time Frame: 6 Weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group
Number analyzed (Participants) | 7 | 4
score on a scale | 40.3 (2.1) | 41.9 (2.3)

3. Secondary Outcome: Effect of Astaxanthin on PROMIS Pain Interference Scores in Patients With Osteoarthritis Who Are Scheduled to Undergo a Total Knee Replacement Surgery.
Description: Patient reported outcomes will be collected utilizing the Patient Reported Outcome Measurement Information Systems (PROMIS) Pain Interference assessment tool. Patients receiving either astaxanthin or placebo will complete the PROMIS Pain Interference assessment prior to starting the oral treatment regimen and just prior to surgery, following the completion of the oral treatment regimen. As the PROMIS tool has national normative data for age, sex, and condition, collection of patient-reported outcomes in this manner will allow for comparison between patients receiving astaxanthin and patients receiving the placebo as well as the general population. A decreased PROMIS Pain Interference score indicates an improvement in patient-reported pain interference. The scale range is 0 to 100 with a mean of 50 and a standard deviation of 10. Higher values are associated with more or higher pain. A score of 60 is one SD worse pain than average. A score of 40 is one SD better pain than average.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group
Number analyzed (Participants) | 7 | 4
score on a scale | 62.0 (2.2) | 55.0 (2.1)

ADVERSE EVENTS:
Time Frame: During study period (approximately one year)
Arm/Group | Control: Placebo Group | Experimental: Astaxanthin Supplementation Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Placebo Group (N=10) | Experimental: Astaxanthin Supplementation Group (N=6)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 2 (2) — stomach pain and discolored stool
Dizziness (General disorders) | 1 (1) | 0 (0) — Dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT05138549/Prot_SAP_ICF_001.pdf